CLINICAL TRIAL: NCT03582449
Title: Intensive Pharmacovigilance Program for Elaprase (SHP ELA-701)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP ELA-701
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hunter Syndrome
Keywords: Hunter syndrome (Mucopolysaccharydosis II)
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elaprase: Participants with Hunter syndrome (Mucopolysaccharydosis II) being treated with Elaprase will be evaluated for this study.

SUMMARY:
The purpose of this non-interventional, observational study which is conducted in Mexico is to evaluate the safety profile of elaprase (idulsurfase) in participants with hunter syndrome (mucopolysaccharydosis II) being treated with elaprase.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders
* Participants to whom idursulfase (Elaprase) has been prescribed
* Participants with Hunter syndrome
* Participants accepting to participate
* Participants signing the informed consent and privacy notice for handling personal information in: the program Contigo Shire (training, diagnosis, family trees) and the intensive pharmacovigilance study for Elaprase. If the participant is unable to provide legal consent (example: under legal age), the participant's legal guardian must provide consent

Exclusion Criteria:

* Participants withdrawing their consent to continue participating in the non-intervention intensive pharmacovigilance study for Elaprase
* Known hypersensitivity or presence of any contraindication to Elaprase that cannot be controlled by pre-medication
* A physical condition that would not permit intravenous administration of enzyme replacement therapy (ERT)
* Participants enrolled in Shire sponsored Elaprase Registry or any other Shire sponsored Elaprase study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with hunter syndrome (mucopolysaccharydosis II) being treated with elaprase will be evaluated for this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events During Administration of Elaprase | During 12 months of study participation
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that do not necessarily have a causal relationship with this treatment. Incidence of adverse events during administration of elaprase will be reported.
Incidence of Adverse Events According to the System Organ Class and MedDRA Preferred Term | During 12 months of study participation
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that do not necessarily have a causal relationship with this treatment. Incidence of adverse events according to the system organ class and MedDRA preferred term will be reported.
Incidence of Adverse Events 2 months After Early Termination of Elaprase Treatment. | 2 months after early termination of Elaprase treatment
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that do not necessarily have a causal relationship with this treatment. Incidence of adverse events 2 months after early termination of Elaprase treatment will be reported.
Change From Baseline in Height Over One Year Study Period | Baseline, 12 months
  Change in height over one year study period will be assessed.
Change From Baseline in Weight Over One Year Study Period | Baseline, 12 months
  Change in weight over one year study period will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Shire Study Physician, Study Director — Shire
Locations (6):
- Mexico (6):
  - Hospital Pediátrico de Sinaloa, Culiacán Rosales, México
  - IMSS UMAE 25 (INSTITUTO MEXICANO DEL SEGURO SOCIAL UNIDAD MEDICA DE ALTA ESPECIALIDAD No 25), Monterrey, Nuevo León
  - Hospital del Niño Tabasqueño, Villahermosa, Tabasco
  - Hospital Centenario Miguel Hidalgo, Aguascalientes
  - Hospital Universitario de Colima, Colima
  - Hospital Infantil Federico Gomez, Mexico City

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual participants could be re-identified (due to the limited number of study participants)

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd24db2bf003ab46ab5